CLINICAL TRIAL: NCT00530777
Title: HSV-2 Suppression to Reduce Maternal HIV-1 RNA Levels During Pregnancy and Breastfeeding
Acronym: VIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Royalty Research Fund - University of Washington (Other); Puget Sound Partners for Global Health (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carey Farquhar, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32462; 07-7306-A01; R03HD057773 (NIH)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: HIV Infections; Herpes Simplex
Keywords: Disease Transmission, Vertical; valacyclovir; Randomized Controlled Trials; HIV; herpes; Herpesvirus 2, Human; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Herpes Simplex | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 500 mg oral valacyclovir twice daily from 34 weeks gestation to 1 year postpartum
  Interventions: Drug: valacyclovir
- 2 (Placebo Comparator): oral placebo twice daily from 34 weeks gestation to 1 year postpartum
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: valacyclovir — 500 mg oral valacyclovir twice daily from 34 weeks gestation to 1 year postpartum
  Other Names: Valtrex
  Arms: 1
Drug: placebo — oral placebo twice daily from 34 weeks gestation to 1 year postpartum
  Arms: 2

SUMMARY:
In this study, we will determine whether treating pregnant and breastfeeding women co-infected with human immunodeficiency virus type 1 (HIV-1) and herpes simplex virus type 2 (HSV-2) with daily valacyclovir will reduce HIV-1 levels in plasma, genital, and breast milk and will decrease the risk of mother-to-child HIV-1 transmission (MTCT).

DETAILED DESCRIPTION:
Each year over 500,000 children become HIV-1-infected in sub-Saharan Africa after exposure to maternal virus in blood, genital secretions, and breast milk. Identifying feasible, safe, and affordable interventions that prevent mother-to-child transmission remains a priority for HIV-1 prevention research. Interventions to reduce breast milk HIV-1 transmission are lacking and most urgently needed.

We propose a randomized clinical trial to determine whether incorporating HSV-2 suppression with valacyclovir into standard prevention of mother-to-child HIV-1 transmission regimens will reduce plasma, cervical, and breast milk HIV-1 RNA levels and risk of transmission among HIV-1-infected and HSV-2-seropositive women. We plan to enroll a total of 148 HIV-1 and HSV-2 co-infected pregnant women with CD4>200 cells/μl who seek antenatal care prior to 32 weeks gestation at a clinic in Nairobi, Kenya. Women will be randomized to receive either valacyclovir suppressive therapy or placebo at 34 weeks gestation and mother-infant pairs will be followed for 12 months postpartum. Follow-up visits will be scheduled at 38 weeks gestation; birth; 2, 6, 10 and 14 weeks; and 6, 9, and 12 months postpartum. Maternal blood, genital, and breast milk specimens obtained at follow-up visits will be used to determine the effect of valacyclovir suppressive therapy on plasma and breast milk HIV-1 RNA levels. Infant filter paper specimens for HIV-1 DNA assays will be collected at birth; 2, 6, 10 and 14 weeks; and 6, 9, and 12 months in order to compare the proportion of infants acquiring HIV-1 by 12 months in the two study arms and determine the timing of HIV-1 infection. In addition, we will monitor maternal and infant renal function in preparation for a larger randomized clinical trial in Africa. The results of this study will help guide the design of a multi-site clinical trial with adequate power to determine the effect of HSV-2 suppression on vertical (MTCT) transmission of HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive
* HSV-2 seropositive
* Plans to deliver in Nairobi
* Resides and plans to remain in Nairobi for 12 months postpartum
* 18 years of age or older
* CD4 count>250 cells/μl

Exclusion Criteria:

* indication for highly active antiretroviral therapy (e.g., WHO stage III or IV)
* hypersensitivity to valacyclovir or acyclovir

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carey Farquhar, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Mathare North City Clinic, Nairobi, Kenya

REFERENCES:
- [Background] Dabis F, Msellati P, Meda N, Welffens-Ekra C, You B, Manigart O, Leroy V, Simonon A, Cartoux M, Combe P, Ouangre A, Ramon R, Ky-Zerbo O, Montcho C, Salamon R, Rouzioux C, Van de Perre P, Mandelbrot L. 6-month efficacy, tolerance, and acceptability of a short regimen of oral zidovudine to reduce vertical transmission of HIV in breastfed children in Cote d'Ivoire and Burkina Faso: a double-blind placebo-controlled multicentre trial. DITRAME Study Group. DIminution de la Transmission Mere-Enfant. Lancet. 1999 Mar 6;353(9155):786-92. doi: 10.1016/s0140-6736(98)11046-2. PMID 10459959
- [Background] Iliff PJ, Piwoz EG, Tavengwa NV, Zunguza CD, Marinda ET, Nathoo KJ, Moulton LH, Ward BJ, Humphrey JH; ZVITAMBO study group. Early exclusive breastfeeding reduces the risk of postnatal HIV-1 transmission and increases HIV-free survival. AIDS. 2005 Apr 29;19(7):699-708. doi: 10.1097/01.aids.0000166093.16446.c9. PMID 15821396
- [Background] Drake AL, John-Stewart GC, Wald A, Mbori-Ngacha DA, Bosire R, Wamalwa DC, Lohman-Payne BL, Ashley-Morrow R, Corey L, Farquhar C. Herpes simplex virus type 2 and risk of intrapartum human immunodeficiency virus transmission. Obstet Gynecol. 2007 Feb;109(2 Pt 1):403-9. doi: 10.1097/01.AOG.0000251511.27725.5c. PMID 17267842
- [Background] Chen KT, Segu M, Lumey LH, Kuhn L, Carter RJ, Bulterys M, Abrams EJ; New York City Perinatal AIDS Collaborative Transmission Study (PACTS) Group. Genital herpes simplex virus infection and perinatal transmission of human immunodeficiency virus. Obstet Gynecol. 2005 Dec;106(6):1341-8. doi: 10.1097/01.AOG.0000185917.90004.7c. PMID 16319261
- [Background] Whitehead S, Bollen L, Leelawiwat W, et al. Maternal HSV-2 Cervicovaginal Shedding Increases the Risk of Intra-partum HIV-1 Transmission. 14th Conference on Retroviruses and Opportunistic Infections. Los Angeles, 2007.
- [Background] Duffus WA, Mermin J, Bunnell R, Byers RH, Odongo G, Ekwaru P, Downing R. Chronic herpes simplex virus type-2 infection and HIV viral load. Int J STD AIDS. 2005 Nov;16(11):733-5. doi: 10.1258/095646205774763298. PMID 16303067
- [Background] Mole L, Ripich S, Margolis D, Holodniy M. The impact of active herpes simplex virus infection on human immunodeficiency virus load. J Infect Dis. 1997 Sep;176(3):766-70. doi: 10.1086/517297. PMID 9291329
- [Background] Mofenson LM, Lambert JS, Stiehm ER, Bethel J, Meyer WA 3rd, Whitehouse J, Moye J Jr, Reichelderfer P, Harris DR, Fowler MG, Mathieson BJ, Nemo GJ. Risk factors for perinatal transmission of human immunodeficiency virus type 1 in women treated with zidovudine. Pediatric AIDS Clinical Trials Group Study 185 Team. N Engl J Med. 1999 Aug 5;341(6):385-93. doi: 10.1056/NEJM199908053410601. PMID 10432323
- [Background] Garcia PM, Kalish LA, Pitt J, Minkoff H, Quinn TC, Burchett SK, Kornegay J, Jackson B, Moye J, Hanson C, Zorrilla C, Lew JF. Maternal levels of plasma human immunodeficiency virus type 1 RNA and the risk of perinatal transmission. Women and Infants Transmission Study Group. N Engl J Med. 1999 Aug 5;341(6):394-402. doi: 10.1056/NEJM199908053410602. PMID 10432324
- [Background] Shaffer N, Roongpisuthipong A, Siriwasin W, Chotpitayasunondh T, Chearskul S, Young NL, Parekh B, Mock PA, Bhadrakom C, Chinayon P, Kalish ML, Phillips SK, Granade TC, Subbarao S, Weniger BG, Mastro TD. Maternal virus load and perinatal human immunodeficiency virus type 1 subtype E transmission, Thailand. Bangkok Collaborative Perinatal HIV Transmission Study Group. J Infect Dis. 1999 Mar;179(3):590-9. doi: 10.1086/314641. PMID 9952365
- [Background] Chuachoowong R, Shaffer N, Siriwasin W, Chaisilwattana P, Young NL, Mock PA, Chearskul S, Waranawat N, Chaowanachan T, Karon J, Simonds RJ, Mastro TD. Short-course antenatal zidovudine reduces both cervicovaginal human immunodeficiency virus type 1 RNA levels and risk of perinatal transmission. Bangkok Collaborative Perinatal HIV Transmission Study Group. J Infect Dis. 2000 Jan;181(1):99-106. doi: 10.1086/315179. PMID 10608756
- [Background] Newell ML. Mechanisms and timing of mother-to-child transmission of HIV-1. AIDS. 1998 May 28;12(8):831-7. doi: 10.1097/00002030-199808000-00004. No abstract available. PMID 9631135
- [Background] Nagot N, Ouedraogo A, Foulongne V, Konate I, Weiss HA, Vergne L, Defer MC, Djagbare D, Sanon A, Andonaba JB, Becquart P, Segondy M, Vallo R, Sawadogo A, Van de Perre P, Mayaud P; ANRS 1285 Study Group. Reduction of HIV-1 RNA levels with therapy to suppress herpes simplex virus. N Engl J Med. 2007 Feb 22;356(8):790-9. doi: 10.1056/NEJMoa062607. PMID 17314338
- [Background] Ozouaki F, Ndjoyi-Mbiguino A, Legoff J, Onas IN, Kendjo E, Si-Mohamed A, Mbopi-Keou FX, Malkin JE, Belec L. Genital shedding of herpes simplex virus type 2 in childbearing-aged and pregnant women living in Gabon. Int J STD AIDS. 2006 Feb;17(2):124-7. doi: 10.1258/095646206775455711. PMID 16464276
- [Background] Conant MA, Schacker TW, Murphy RL, Gold J, Crutchfield LT, Crooks RJ; International Valaciclovir HSV Study Group. Valaciclovir versus aciclovir for herpes simplex virus infection in HIV-infected individuals: two randomized trials. Int J STD AIDS. 2002 Jan;13(1):12-21. doi: 10.1258/0956462021924550. PMID 11802924
- [Background] Workowski KA, Berman SM. Centers for Disease Control and Prevention sexually transmitted diseases treatment guidelines. Clin Infect Dis. 2007 Apr 1;44 Suppl 3:S73-6. doi: 10.1086/511430. No abstract available. PMID 17342670
- [Background] Sheffield JS, Hill JB, Hollier LM, Laibl VR, Roberts SW, Sanchez PJ, Wendel GD Jr. Valacyclovir prophylaxis to prevent recurrent herpes at delivery: a randomized clinical trial. Obstet Gynecol. 2006 Jul;108(1):141-7. doi: 10.1097/01.AOG.0000219749.96274.15. PMID 16816068
- [Background] Andrews WW, Kimberlin DF, Whitley R, Cliver S, Ramsey PS, Deeter R. Valacyclovir therapy to reduce recurrent genital herpes in pregnant women. Am J Obstet Gynecol. 2006 Mar;194(3):774-81. doi: 10.1016/j.ajog.2005.11.051. PMID 16522412
- [Background] Kimberlin DF, Weller S, Whitley RJ, Andrews WW, Hauth JC, Lakeman F, Miller G. Pharmacokinetics of oral valacyclovir and acyclovir in late pregnancy. Am J Obstet Gynecol. 1998 Oct;179(4):846-51. doi: 10.1016/s0002-9378(98)70176-0. PMID 9790357
- [Background] Ashley RL, Militoni J, Lee F, Nahmias A, Corey L. Comparison of Western blot (immunoblot) and glycoprotein G-specific immunodot enzyme assay for detecting antibodies to herpes simplex virus types 1 and 2 in human sera. J Clin Microbiol. 1988 Apr;26(4):662-7. doi: 10.1128/jcm.26.4.662-667.1988. PMID 2835389
- [Background] Panteleeff DD, John G, Nduati R, Mbori-Ngacha D, Richardson B, Kreiss J, Overbaugh J. Rapid method for screening dried blood samples on filter paper for human immunodeficiency virus type 1 DNA. J Clin Microbiol. 1999 Feb;37(2):350-3. doi: 10.1128/JCM.37.2.350-353.1999. PMID 9889216
- [Derived] Roxby AC, Atkinson C, Asbjornsdottir K, Farquhar C, Kiarie JN, Drake AL, Wald A, Boeckh M, Richardson B, Emery V, John-Stewart G, Slyker JA. Maternal valacyclovir and infant cytomegalovirus acquisition: a randomized controlled trial among HIV-infected women. PLoS One. 2014 Feb 4;9(2):e87855. doi: 10.1371/journal.pone.0087855. eCollection 2014. PMID 24504006
- [Derived] Roxby AC, Liu AY, Drake AL, Kiarie JN, Richardson B, Lohman-Payne BL, John-Stewart GC, Wald A, De Rosa S, Farquhar C. Short communication: T cell activation in HIV-1/herpes simplex virus-2-coinfected Kenyan women receiving valacyclovir. AIDS Res Hum Retroviruses. 2013 Jan;29(1):94-8. doi: 10.1089/AID.2012.0071. Epub 2012 Sep 4. PMID 22852760
- [Derived] Drake AL, Roxby AC, Kiarie J, Richardson BA, Wald A, John-Stewart G, Farquhar C. Infant safety during and after maternal valacyclovir therapy in conjunction with antiretroviral HIV-1 prophylaxis in a randomized clinical trial. PLoS One. 2012;7(4):e34635. doi: 10.1371/journal.pone.0034635. Epub 2012 Apr 11. PMID 22509337
- [Derived] Drake AL, Roxby AC, Ongecha-Owuor F, Kiarie J, John-Stewart G, Wald A, Richardson BA, Hitti J, Overbaugh J, Emery S, Farquhar C. Valacyclovir suppressive therapy reduces plasma and breast milk HIV-1 RNA levels during pregnancy and postpartum: a randomized trial. J Infect Dis. 2012 Feb 1;205(3):366-75. doi: 10.1093/infdis/jir766. Epub 2011 Dec 6. PMID 22147786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-1 infected pregnant women seeking antenatal care at the Mathare North City Council Clinic in Nairobi Kenya, or referred from neighboring clinics, were recruited for study screening
Period: Overall Study
Arm/Group | Valacyclovir | Placebo
Started | 74 | 74
Completed | 67 | 69
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unable to adhere to visit schedule | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 71 | 70 | 141
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.3) | 26.0 (4.5) | 26.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 74 | 74 | 148

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HIV-1 Levels in Plasma Between 34 and 38 Weeks Gestation
Description: Calculated as log10 plasma viral load at 34 weeks gestation - log10 plasma viral load at 38 weeks gestation
Time Frame: 4 weeks
Population: Women with paired plasma samples at 34 and 38 weeks gestation
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 51 | 49
log10 copies/mL | -0.53 (.074) | 0.03 (0.76)

2. Secondary Outcome: Vertical HIV-1 Transmission
Description: Mother-to-child HIV transmission
Time Frame: 1 year postpartum
Population: Note the sample size is 73 for each group rather than 74 due to loss to follow-up.
Measure: Number; unit: Participants
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 73 | 73
Participants | 6 | 4

ADVERSE EVENTS:
Arm/Group | Valacyclovir | Placebo
Serious Adverse Events (participants affected / at risk) | 1/74 | 2/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Valacyclovir (N=74) | Placebo (N=74)
Death (Investigations) | 1/1 (1) | 2/2 (2)

LIMITATIONS AND CAVEATS:
Unable to evaluate the effect of valacyclovir on mother-to-child HIV transmission (MTCT) or on change in HIV-1 RNA among women eligible for highly active antiretroviral therapy (HAART); lack power to detect association between treatment and MTCT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No